CLINICAL TRIAL: NCT04816760
Title: Alterations of Innate and Adaptive Immune Cells During the Course of SARS CoV-2 Pneumonia
Brief Title: Immune Cells Phenotypes During COVID-19
Acronym: IMMUNO-COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Hospitalo-Universitaire Méditerranée Infection (Other)
Collaborators: Hôpital Européen Marseille (Other); Assistance Publique Hopitaux De Marseille (Other); Institut Paoli-Calmettes (Other); Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-A00756-33
Record Dates: First submitted 2021-02-12; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Sars-CoV2; Innate Immunity; Immunization; Infection; Alveolar Lung Disease; Endothelial Dysfunction
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Peripheral blood samples — Peripheral blood samples at Day 0, Day 7, Day 14, Day 28, Day 90 and Day 180.

SUMMARY:
The ongoing pandemic caused by the Severe Acute Respiratory Syndrome Coronavirus 2 (SARS CoV-2) has infected more than one hundred twenty million peoples worldwide one year after its onset with a case-fatality rate of almost 2%. The disease due to the coronavirus 2019 (i.e., COVID-19) is associated with a wide range of clinical symptoms. As the primary site of viral invasion is the upper respiratory airways, lung infection is the most common complication. Most infected patients are asymptomatic or experience mild or moderate form of the disease (80 %). A lower proportion (15%) develop severe pneumonia with variable level of hypoxia that may required hospitalization for oxygen therapy. In the most severe cases (5%), patients evolve towards critical illness with organ failure such as the acute respiratory distress syndrome (ARDS). At this stage, invasive mechanical ventilation is required in almost 70 % and the hospital mortality rises to 37 %.

Immune cells are key players during SARS CoV-2 infection and several alterations have been reported including lymphocytes (T, B and NK) and monocytes depletion, and cells exhaustion. Such alterations were much more pronounced in patients with the most severe form of the disease. Beside, a dysregulated proinflammatory response has also been pointed out as a potential mechanism of lung damage. Finally, COVID-19 is associated with an unexpectedly high incidence of thrombosis which probably results from the viral invasion of endothelial cells.

The investigators aim to explore prospectively the alterations of innate and adaptive immune cells during both the acute and the recovery phase of SARS CoV-2 pneumonia. Flow and Spectral cytometry will be used to perform deep subset profiling focusing on T, B, NK, NKT, gamma-gelta T, monocytes and dendritic cells. Each specific cell type will be further characterized using markers of activation/inhibition, maturation/differenciation and senescence as well as chemokines receptors.

T-cell memory specificity will be explore using specific SARS CoV-2 pentamer. Platelet activation and circulating microparticles will be explore using flow cytometry. Serum SARS CoV-2 antibodies (IgA, IgM, IgG), serum cytokines, and serum biomarkers of alveolar epithelial and endothelial cells will be analyze using ELISA and correlate with the severity of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 y
* Laboratory confirmed SARS CoV-2 infection (positive RT-PCR).
* Ground-glass opacity on chest computed-tomography
* Time from hospital admission to inclusion < or equal to 72 h

Exclusion Criteria:

* Pregnant
* Under legal restriction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting with a first episode of SARS CoV-2 pneumonia and requiring hospitalization either in a ward or an Intensive Care Unit will constitute the COVID-19 group.
  Healthy blood donors from the Etablissement Français du Sang (EFS) will constituted the control group
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-25 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Profiling of innate and adaptive immune cells during SARS CoV-2 infection. | Day 0
  Determination of cells population using spectral cytometry of PBMCs.
Profiling of innate and adaptive immune cells during SARS CoV-2 infection. | Day 7
  Determination of cells population using spectral cytometry of PBMCs.
Profiling of innate and adaptive immune cells during SARS CoV-2 infection. | Day 14
  Determination of cells population using spectral cytometry of PBMCs.
Profiling of innate and adaptive immune cells during SARS CoV-2 infection. | Day 28
  Determination of cells population using spectral cytometry of PBMCs.
Profiling of innate and adaptive immune cells during SARS CoV-2 infection. | Day 90
  Determination of cells population using spectral cytometry of PBMCs.
Profiling of innate and adaptive immune cells during SARS CoV-2 infection. | Day 180
  Determination of cells population using spectral cytometry of PBMCs.
Functional state of innate and adaptive immune cells during SARS CoV-2 infection. | Day 0
  Determination of the functional state of immune cells using spectral cytometry
Functional state of innate and adaptive immune cells during SARS CoV-2 infection. | Day 7
  Determination of the functional state of immune cells using spectral cytometry
Functional state of innate and adaptive immune cells during SARS CoV-2 infection. | Day 14
  Determination of the functional state of immune cells using spectral cytometry
Functional state of innate and adaptive immune cells during SARS CoV-2 infection. | Day 28
  Determination of the functional state of immune cells using spectral cytometry
Functional state of innate and adaptive immune cells during SARS CoV-2 infection. | Day 90
  Determination of the functional state of immune cells using spectral cytometry
Functional state of innate and adaptive immune cells during SARS CoV-2 infection. | Day 180
  Determination of the functional state of immune cells using spectral cytometry
Serum IgA, IgM and IgG antibodies during SARS CoV-2 infection. | Day 0
  Measurement of serum SARS CoV-2 IgA, IgM and IgG antibodies using Elisa.
Serum IgA, IgM and IgG antibodies during SARS CoV-2 infection. | Day 7
  Measurement of serum SARS CoV-2 IgA, IgM and IgG antibodies using Elisa.
Serum IgA, IgM and IgG antibodies during SARS CoV-2 infection. | Day 14
  Measurement of serum SARS CoV-2 IgA, IgM and IgG antibodies using Elisa.
Serum IgA, IgM and IgG antibodies during SARS CoV-2 infection. | Day 28
  Measurement of serum SARS CoV-2 IgA, IgM and IgG antibodies using Elisa.
Serum IgA, IgM and IgG antibodies during SARS CoV-2 infection. | Day 90
  Measurement of serum SARS CoV-2 IgA, IgM and IgG antibodies using Elisa.
Serum IgA, IgM and IgG antibodies during SARS CoV-2 infection. | Day 180
  Measurement of serum SARS CoV-2 IgA, IgM and IgG antibodies using Elisa.
Platelet activation and circulating microparticles assessment during SARS CoV-2 infection. | Day 0
  Determination of platelet activation and circulating microparticles levels using flow cytometry.
Platelet activation and circulating microparticles assessment during SARS CoV-2 infection. | Day 7
  Determination of platelet activation and circulating microparticles levels using flow cytometry.
Platelet activation and circulating microparticles assessment during SARS CoV-2 infection. | Day 14
  Determination of platelet activation and circulating microparticles levels using flow cytometry.
Platelet activation and circulating microparticles assessment during SARS CoV-2 infection. | Day 28
  Determination of platelet activation and circulating microparticles levels using flow cytometry.

SECONDARY OUTCOMES:
Serum concentration of Pro-inflammatory and Anti-inflammatory cytokines in response to SARS CoV-2 infection. | Day 0
  Measurement of IL1β, IL-6, IL-10, IL-17A, IL-18, TNFα, IFNγ, CRTP-6 using Elisa.
Serum concentration of Pro-inflammatory and Anti-inflammatory cytokines in response to SARS CoV-2 infection. | Day 7
  Measurement of IL1β, IL-6, IL-10, IL-17A, IL-18, TNFα, IFNγ, CRTP-6 using Elisa.
Serum concentration of Pro-inflammatory and Anti-inflammatory cytokines in response to SARS CoV-2 infection. | Day 14
  Measurement of IL1β, IL-6, IL-10, IL-17A, IL-18, TNFα, IFNγ, CRTP-6 using Elisa.
Serum concentration of Pro-inflammatory and Anti-inflammatory cytokines in response to SARS CoV-2 infection. | Day 28
  Measurement of IL1β, IL-6, IL-10, IL-17A, IL-18, TNFα, IFNγ, CRTP-6 using Elisa.
Serum concentration of Pro-inflammatory and Anti-inflammatory cytokines in response to SARS CoV-2 infection. | Day 90
  Measurement of IL1β, IL-6, IL-10, IL-17A, IL-18, TNFα, IFNγ, CRTP-6 using Elisa.
Serum concentration of Pro-inflammatory and Anti-inflammatory cytokines in response to SARS CoV-2 infection. | Day 180
  Measurement of IL1β, IL-6, IL-10, IL-17A, IL-18, TNFα, IFNγ, CRTP-6 using Elisa.
Serum alveolar epithelial and endothelial cells biomarkers during SARS CoV-2 infection. | Day 0
  Measurement of KL-6, CC-16, S-RAGE, ANG-2 using ELISA.
Serum alveolar epithelial and endothelial cells biomarkers during SARS CoV-2 infection. | Day 7
  Measurement of KL-6, CC-16, S-RAGE, ANG-2 using ELISA.
Serum alveolar epithelial and endothelial cells biomarkers during SARS CoV-2 infection. | Day 14
  Measurement of KL-6, CC-16, S-RAGE, ANG-2 using ELISA.
Serum alveolar epithelial and endothelial cells biomarkers during SARS CoV-2 infection. | Day 28
  Measurement of KL-6, CC-16, S-RAGE, ANG-2 using ELISA.
Kinetic of surface biomarkers expression on neutrophils (C64) and monocytes (CD169, HLA-DR) during SARS CoV-2 infection. | Day 0
  Measurement of nCD64, mCD169 and mHLA-DR using the VersaPOC one-step rapid flow cytometry method.
Kinetic of surface biomarkers expression on neutrophils (C64) and monocytes (CD169, HLA-DR) during SARS CoV-2 infection. | Day 1
  Measurement of nCD64, mCD169 and mHLA-DR using the VersaPOC one-step rapid flow cytometry method.
Kinetic of surface biomarkers expression on neutrophils (C64) and monocytes (CD169, HLA-DR) during SARS CoV-2 infection. | Day 2
  Measurement of nCD64, mCD169 and mHLA-DR using the VersaPOC one-step rapid flow cytometry method.
Kinetic of surface biomarkers expression on neutrophils (C64) and monocytes (CD169, HLA-DR) during SARS CoV-2 infection. | Day 3
  Measurement of nCD64, mCD169 and mHLA-DR using the VersaPOC one-step rapid flow cytometry method.
Kinetic of surface biomarkers expression on neutrophils (C64) and monocytes (CD169, HLA-DR) during SARS CoV-2 infection. | Day 5
  Measurement of nCD64, mCD169 and mHLA-DR using the VersaPOC one-step rapid flow cytometry method.
Kinetic of surface biomarkers expression on neutrophils (C64) and monocytes (CD169, HLA-DR) during SARS CoV-2 infection. | Day 7
  Measurement of nCD64, mCD169 and mHLA-DR using the VersaPOC one-step rapid flow cytometry method.
Kinetic of surface biomarkers expression on neutrophils (C64) and monocytes (CD169, HLA-DR) during SARS CoV-2 infection. | Day 9
  Measurement of nCD64, mCD169 and mHLA-DR using the VersaPOC one-step rapid flow cytometry method.
Kinetic of surface biomarkers expression on neutrophils (C64) and monocytes (CD169, HLA-DR) during SARS CoV-2 infection. | Day 11
  Measurement of nCD64, mCD169 and mHLA-DR using the VersaPOC one-step rapid flow cytometry method.
Kinetic of surface biomarkers expression on neutrophils (C64) and monocytes (CD169, HLA-DR) during SARS CoV-2 infection. | Day 14
  Measurement of nCD64, mCD169 and mHLA-DR using the VersaPOC one-step rapid flow cytometry method.
Kinetic of surface biomarkers expression on neutrophils (C64) and monocytes (CD169, HLA-DR) during SARS CoV-2 infection. | Day 17
  Measurement of nCD64, mCD169 and mHLA-DR using the VersaPOC one-step rapid flow cytometry method.
Kinetic of surface biomarkers expression on neutrophils (C64) and monocytes (CD169, HLA-DR) during SARS CoV-2 infection. | Day 21
  Measurement of nCD64, mCD169 and mHLA-DR using the VersaPOC one-step rapid flow cytometry method.
Kinetic of surface biomarkers expression on neutrophils (C64) and monocytes (CD169, HLA-DR) during SARS CoV-2 infection. | Day 28
  Measurement of nCD64, mCD169 and mHLA-DR using the VersaPOC one-step rapid flow cytometry method.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis MEGE, MD, PhD, Principal Investigator — Institut Hospitalo-Universitaire Méditérranée Infection
Locations (2):
- France (2):
  - Hopital Europeen Marseille, Marseille
  - Hopital Nord, Marseille

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Kuri-Cervantes L, Pampena MB, Meng W, Rosenfeld AM, Ittner CAG, Weisman AR, Agyekum RS, Mathew D, Baxter AE, Vella LA, Kuthuru O, Apostolidis SA, Bershaw L, Dougherty J, Greenplate AR, Pattekar A, Kim J, Han N, Gouma S, Weirick ME, Arevalo CP, Bolton MJ, Goodwin EC, Anderson EM, Hensley SE, Jones TK, Mangalmurti NS, Luning Prak ET, Wherry EJ, Meyer NJ, Betts MR. Comprehensive mapping of immune perturbations associated with severe COVID-19. Sci Immunol. 2020 Jul 15;5(49):eabd7114. doi: 10.1126/sciimmunol.abd7114. PMID 32669287
- [Background] Giamarellos-Bourboulis EJ, Netea MG, Rovina N, Akinosoglou K, Antoniadou A, Antonakos N, Damoraki G, Gkavogianni T, Adami ME, Katsaounou P, Ntaganou M, Kyriakopoulou M, Dimopoulos G, Koutsodimitropoulos I, Velissaris D, Koufargyris P, Karageorgos A, Katrini K, Lekakis V, Lupse M, Kotsaki A, Renieris G, Theodoulou D, Panou V, Koukaki E, Koulouris N, Gogos C, Koutsoukou A. Complex Immune Dysregulation in COVID-19 Patients with Severe Respiratory Failure. Cell Host Microbe. 2020 Jun 10;27(6):992-1000.e3. doi: 10.1016/j.chom.2020.04.009. Epub 2020 Apr 21. PMID 32320677
- [Background] Qin C, Zhou L, Hu Z, Zhang S, Yang S, Tao Y, Xie C, Ma K, Shang K, Wang W, Tian DS. Dysregulation of Immune Response in Patients With Coronavirus 2019 (COVID-19) in Wuhan, China. Clin Infect Dis. 2020 Jul 28;71(15):762-768. doi: 10.1093/cid/ciaa248. PMID 32161940
- [Background] Zheng M, Gao Y, Wang G, Song G, Liu S, Sun D, Xu Y, Tian Z. Functional exhaustion of antiviral lymphocytes in COVID-19 patients. Cell Mol Immunol. 2020 May;17(5):533-535. doi: 10.1038/s41423-020-0402-2. Epub 2020 Mar 19. No abstract available. PMID 32203188
- [Background] Hue S, Beldi-Ferchiou A, Bendib I, Surenaud M, Fourati S, Frapard T, Rivoal S, Razazi K, Carteaux G, Delfau-Larue MH, Mekontso-Dessap A, Audureau E, de Prost N. Uncontrolled Innate and Impaired Adaptive Immune Responses in Patients with COVID-19 Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2020 Dec 1;202(11):1509-1519. doi: 10.1164/rccm.202005-1885OC. PMID 32866033
- [Background] Ackermann M, Verleden SE, Kuehnel M, Haverich A, Welte T, Laenger F, Vanstapel A, Werlein C, Stark H, Tzankov A, Li WW, Li VW, Mentzer SJ, Jonigk D. Pulmonary Vascular Endothelialitis, Thrombosis, and Angiogenesis in Covid-19. N Engl J Med. 2020 Jul 9;383(2):120-128. doi: 10.1056/NEJMoa2015432. Epub 2020 May 21. PMID 32437596
- [Derived] Gay L, Rouviere MS, Mezouar S, Richaud M, Gorvel L, Foucher E, La Scola B, Menard A, Allardet-Servent J, Halfon P, Frohna P, Cano C, Mege JL, Olive D. Vgamma9Vdelta2 T-cells Are Potent Inhibitors of SARS-CoV-2 Replication and Represent Effector Phenotypes in Patients With COVID-19. J Infect Dis. 2024 Jun 14;229(6):1759-1769. doi: 10.1093/infdis/jiae169. PMID 38557809
- See also: WHO Coronavirus Disease (COVID-19) Dashboard — https://covid19.who.int/